CLINICAL TRIAL: NCT03532451
Title: Phase Ib Feasibility Trial of Neoadjuvant Nivolumab/Lirilumab in Cisplatin-Ineligible Muscle-Invasive Bladder Cancer
Acronym: PrE0807
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PrECOG, LLC. (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PrE0807; CA209-9DF (Other: BMS)
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Results first posted 2021-09-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer
Keywords: Muscle-Invasive; Cisplatin-Ineligible; Nivolumab; Lirilumab
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Nivolumab; lirilumab

STUDY DESIGN:
Intervention Model Description: Cohort 1: Nivolumab alone (Completed November 20, 2019). In the absence of the occurrence of high rate of treatment related adverse events, the study will proceed with enrollment into Cohort 2: Nivolumab/Lirilumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Nivolumab (Experimental): Nivolumab 480 mg IV on week 0 and week 4
  Interventions: Drug: Nivolumab
- Cohort 2: Nivolumab/Lirilumab (Experimental): Nivolumab 480 mg IV and Lirilumab 240 mg on week 0 and week 4
  Interventions: Drug: Nivolumab/Lirilumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 480 mg intravenously (IV) over approximately 30 minutes every 4 weeks for 2 neo-adjuvant doses (week 0 and 4) followed by RC with bilateral (standard or extended) PLND as soon as possible but within 6 weeks after the last neoadjuvant infusion.
  Other Names: Opdivo
  Arms: Cohort 1: Nivolumab
Drug: Nivolumab/Lirilumab — Nivolumab 480 mg IV over approximately 60 minutes every 4 weeks for 2 neo-adjuvant doses (week 0 and 4) with at least a 30 minute rest between infusions followed by lirilumab 240 mg IV over approximately 60 minutes every 4 weeks for 2 neo-adjuvant doses (week 0 and 4) followed by RC with bilateral (standard or extended) PLND as soon as possible but within 6 weeks after the last neoadjuvant infusion.
  Other Names: Opdivo; BMS-986015
  Arms: Cohort 2: Nivolumab/Lirilumab

SUMMARY:
Patients with muscle-invasive bladder cancer (MIBC) who can not receive cisplatin or refuse cisplatin therapy will receive nivolumab or nivolumab/lirilumab before a planned surgical procedure called a radical cystectomy (RC) to remove the bladder.

Nivolumab works by attaching to and blocking a molecule called Programmed Death-1 (PD-1). Lirilumab attaches to and blocks a group of molecules called Killer Cell Immunoglobulin-Like Receptor (KIR). PD-1 and KIR are proteins present mainly on immune system cells, and each controls part of the immune system by shutting it down. It is hoped that by binding to and inactivating these proteins, these drugs can enhance the body's ability to detect, attack and destroy cancer cells.

The purpose of this research study is to see whether nivolumab alone or combination of nivolumab and lirilumab given before surgery is effective in treating people who have bladder cancer, and to examine the side effects, good and bad, associated with nivolumab and lirilumab.

DETAILED DESCRIPTION:
Bladder cancer (BC) is the 6th most common malignancy in the United States with an estimated 79,030 new cases and 16,870 deaths in 2017. It is the 4th most common cancer in men and there are presently >500,000 BC patients alive in the US. It accounts for about 5% of all new cancers in the US. It is also the most expensive cancer to treat from diagnosis to death. Almost a third of BC patients present with MIBC.

This is a Phase Ib open-label clinical trial for patients that are either cisplatin-ineligible or refuse cisplatin-based chemotherapy and have MIBC (T2-T4a, N0-N1, M0).Neoadjuvant treatment must start within 10 weeks of transurethral resection of the most recent transurethral resection of bladder tumor (TURBT) that showed muscularis propria invasion.

Patients must have sufficient baseline tumor tissue. Tumor tissue content for CD8+ T-cell density assessment must be qualified as sufficient (≥ 20% tumor content in the specimen) for analysis and must be documented by the local pathologist prior to registration.

The first 12 patients will be enrolled into Cohort 1 and treated with nivolumab before a planned RC (Completed November 20, 2019).

In the absence of the occurrence of high rate of treatment related Adverse Events (AEs) with nivolumab, the study will proceed with enrollment into Cohort 2 with the combination of nivolumab/lirilumab before a planned RC.

Each group will receive a total of 2 doses (week 0 and 4) of nivolumab (Cohort 1) or nivolumab/lirilumab (Cohort 2) therapy followed by RC with bilateral (standard or extended) pelvic lymph node dissection (PLND).

Mandatory tumor tissue at Screening (archived tumor tissue from Transurethral Resection of Bladder Tumor [TURBT] may be used) and at time of RC. Peripheral blood and urine samples are also required.

ELIGIBILITY:
* Patients must have histologically confirmed MIBC (T2-T4a, N0-N1, M0 per American Joint Commission on Cancer [AJCC]) pure or mixed histology urothelial carcinoma. Clinical node-positive (N1) patients are eligible provided the lymph nodes (LNs) are confined to the true pelvis and are within the planned surgical LN dissection template.
* The most recent TURBT that showed muscularis propria invasion should be within 10 weeks prior to beginning study therapy. Patients must have sufficient baseline tumor tissue from either initial or repeat TURBTs. The local site pathologist will be asked to estimate and record the rough approximate percentage of viable tumor in the TURBT sample (initial or repeat TURBT with highest tumor content) to document at least 20% viable tumor content prior to registration.
* Patients must be ineligible for cisplatin-based chemotherapy due to any of the following below OR refused cisplatin-based chemotherapy:

  * Creatinine clearance(CrCl) <60 mL/min with Easter Cooperative Oncology Group (ECOG) Performance Status (PS) 0-1
  * Creatinine clearance(CrCl) ≥ 60 mL/min with ECOG PS 2 (if patient fit for RC)
  * Hearing impaired ≥ Grade 2 by CTCAE criteria
  * Neuropathy ≥ Grade 2 by CTCAE criteria
  * Patient refused cisplatin-based chemotherapy?
* Patients must be medically fit for TURBT and RC.
* Age ≥ 18 years.
* Ability to understand and willingness to sign Institutional Review Board (IRB)-approved informed consent.
* Willing to provide tumor tissue, blood, and urine samples for research.
* Adequate organ function as measured by the following criteria, obtained ≤ 4 weeks prior to registration:

  * Absolute Neutrophil Count (ANC) ≥ 1000/mm³ (stable off growth factor within 4 weeks of first study drug administration)
  * Platelets ≥ 100,000/mm³
  * Hemoglobin ≥ 8 g/dL
  * Serum Creatinine Clearance ≥ 30 mL/min using the Cockcroft-Gault formula
  * Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) ≤ 3x Upper Limit of Normal (ULN)
  * Total Bilirubin ≤ 1.5x ULN (in the absence of previously diagnosed Gilbert's disease)
* Women must not be pregnant or breastfeeding since we do not know the effects of nivolumab and lirilumab on the fetus or breastfeeding child.
* Sexually active women of child-bearing potential with a non-sterilized male partner and sexually active men must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) OR abstinence prior to study entry, for the duration of study participation, and for 5 months for women and 7 months for men following last dose of study drugs.
* Active or prior documented autoimmune disease within the past 2 years prior to Screening or other immunosuppressive agent within 14 days of study treatment.
* Patients may not have locally advanced unresectable or metastatic urothelial carcinoma as assessed on baseline radiographic imaging obtained within 28 days prior to study registration.
* Patients may not have concurrent upper urinary tract (i.e. ureter, renal pelvis) invasive urothelial carcinoma. Patients with history of non-invasive (Ta, Tis) upper tract urothelial carcinoma that has been definitively treated with at least one post-treatment disease assessment (i.e. cytology, biopsy, imaging) that demonstrates no evidence of residual disease are eligible.
* Patients may not have another malignancy that could interfere with the evaluation of safety or efficacy of the study drugs. Patients with a prior malignancy will be allowed without study chair approval in the following circumstances:

  * Not currently active and diagnosed at least 3 years prior to the date of registration.
  * Non-invasive diseases such as low risk cervical cancer or any cancer in situ.
  * Localized (early stage) cancer treated with curative intent (without evidence of recurrence and intent for further therapy), and in which no systemic chemotherapy was indicated.(e.g. low/intermediate risk prostate cancer, etc.).
* Patients may not have received any prior immune checkpoint inhibitor (i.e. anti-KIR, anti-PD-1, anti-PD-L1, or other).
* Patients may not have undergone major surgery (e.g. intra-thoracic, intra-abdominal or intra-pelvic), open biopsy or significant traumatic injury or specific anti-cancer treatment ≤ 4 weeks prior to starting study drug, or patients who have had percutaneous biopsies or placement of vascular access device ≤ 1 week prior to starting study drug, or who have not recovered from side effects of such procedure or injury.
* Patients must not have clinically significant cardiac disease.
* Patients may not have chronic active liver disease or evidence of acute or chronic Hepatitis B Virus (HBV) or Hepatitis C (HCV).
* Patients may not have known diagnosis of human immunodeficiency virus (HIV) infection. Testing is not required in absence of clinical suspicion.
* Patients may not have known diagnosis of any condition (e.g. post-hematopoietic or solid visceral organ transplant, pneumonitis, inflammatory bowel disease, etc.) that requires chronic immunosuppressive therapy. Usage of non-steroidal anti-inflammatory medications (NSAIDS) for the treatment of osteoarthritis and uric acid synthesis inhibitors for the treatment of gout are permitted.
* Patients with any serious and/or uncontrolled concurrent medical conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) or psychiatric illness that could, in the investigator's opinion, cause unacceptable safety risks or potentially interfere with the completion of the treatment according to the protocol are not eligible.
* Patients may not have any live viral vaccine used for prevention of infectious diseases within 4 weeks prior to study drug(s).
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petros Grivas, MD, PhD, Study Chair — University of Washington
Locations (8):
- United States (8):
  - Moffitt Cancer Center, Tampa, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of TX Southwestern, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

REFERENCES:
- [Result] Grivas P, Koshkin VS, Chu X, Cole S, Jain RK, Dreicer R, Cetnar JP, Sundi D, Gartrell BA, Galsky MD, Woo B, Li-Ning-Tapia E, Hahn NM, Carducci MA. PrECOG PrE0807: A Phase 1b Feasibility Trial of Neoadjuvant Nivolumab Without and with Lirilumab in Patients with Muscle-invasive Bladder Cancer Ineligible for or Refusing Cisplatin-based Neoadjuvant Chemotherapy. Eur Urol Oncol. 2024 Aug;7(4):914-922. doi: 10.1016/j.euo.2023.11.022. Epub 2023 Dec 27. PMID 38155060

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab
Started | 13 | 30
Completed | 12 | 28
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Did not undergo surgery | 1 | 1

BASELINE CHARACTERISTICS:
Population: One patient was excluded from the reporting of baseline data due to withdrawal consent prior to any treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab | Total
Number analyzed (Participants) | 13 | 29 | 42
Age, Continuous [Median (Full Range); unit: years] | 76 [60 to 89] | 75 [51 to 83] | 75 [51 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 14
  Male | 10 | 18 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 27 | 38
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 13 | 27 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
ECOG Performance Status [Count of Participants; unit: Participants] — 0-Fully active, able to carry on all pre-disease performance without restriction;
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 10 | 18 | 28
    1 | 2 | 11 | 13
    2 | 1 | 0 | 1
Prior Chemotherapy [Count of Participants; unit: Participants] | 2 | 3 | 5
Clinical Stage [Count of Participants; unit: Participants] — Clinical stage of the disease was diagnosed according to CT or MRI in relation to clinical data. Higher numbers mean the cancer is more advanced. The earliest stage cancers are called stage 0 (or carcinoma in situ), and then range from stages I (1) through IV (4) T0. No evidence as primary tumor T1-T4. Size and/or extent of the primary tumor NX. Regional lymph nodes cannot be evaluated N0. No regional lymph node involvement (no cancer found in the lymph nodes) N1-N3. Involvement of regional lymph nodes (number and/or extent of spread)
  Participants
    cT2 N0 | 10 | 23 | 33
    cT3 N0 | 1 | 0 | 1
    cT4 N0 | 1 | 2 | 3
    cT2-4a N1 | 1 | 1 | 2
    cT2-4a Nx | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 or Higher Treatment Related Adverse Events as Assessed by CTCAE V5.0
Description: To assess safety of treatment according to Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) manifested as the rate of Grade 3 or higher treatment related adverse events in patients treated with nivolumab (Cohort 1) or combination of nivolumab/lirilumab (Cohort 2). The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. Toxicity graded by CTCAE v5.0 scaling from 1-5 (mild to death). Grade 3 or higher events are those that are graded '3- severe or medically significant', 4- life-threatening consequences; urgent intervention indicated' or '5-Death related to AE'.
Time Frame: 16 months
Population: Patients who received any treatment.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab
Number analyzed (Participants) | 13 | 29
proportion of participants | 0 [0 to 0.21] | 0.07 [0.01 to 0.20]

2. Secondary Outcome: Percentage of Participants With Pathologic Complete and Partial Response
Description: Measured by pathologic complete (pT0N0) and partial (<pT2N0) response rate at time of RC in the two cohorts
Time Frame: Responses was assessed at baseline and time of radical cystectomy (within 6 weeks after the last treatment), up to 6 months.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab
Number analyzed (Participants) | 12 | 28
percentage of participants
  ypT0N0 | 16.7 [3.0 to 43.8] | 21.4 [9.8 to 38.0]
  <ypT2N0 | 25.0 [7.2 to 52.7] | 32.1 [17.9 to 49.4]

3. Secondary Outcome: Two Year Recurrence-free Survival
Description: Measured by recurrence rate after 2 years following the RC in the two cohorts.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: percentage of RFS patients
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab
Number analyzed (Participants) | 12 | 28
percentage of RFS patients | 82 [61.9 to 100] | 89 [78.5 to 100]

4. Secondary Outcome: Rate of no RC Due to TRAEs
Description: the rate of patients in each cohort who do not get RC within 6 weeks after completion of neoadjuvant treatment specifically and directly related to treatment-related adverse events (AEs)
Time Frame: from completion of neoadjuvant treatment to 6 weeks after
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab
Number analyzed (Participants) | 12 | 28
Participants | 0 | 0

5. Secondary Outcome: Change in CD8+ TIL Density
Description: CD8+ TIL density was measured at baseline(TURBT) and radical cystectomy after treatment. Change in CD8+ TIL density from pre-treatment Transurethral Resection of Bladder Tumor (TURBT) to post-treatment Radical Cystectomy (RC) tissues separately in patients treated with nivolumab or combination of nivolumab/lirilumab. Each individual patient's CD8+ TIL density change was defined as number of CD8+ cells / the annotated tissue area in mm2
Time Frame: From pre-treatment Transurethral Resection of Bladder Tumor (TURBT) which happens 10 weeks (at most) before treatment to post-treatment Radical Cystectomy (RC), up to 6 months. RC was scheduled within 6 weeks after the last neoadjuvant infusion
Measure: Median (Full Range); unit: percent of CD8+ cells
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab
Number analyzed (Participants) | 12 | 28
percent of CD8+ cells | 120.5 [-508.9 to 809.8] | 126.9 [-235.6 to 939.6]
Statistical Analysis 1: Comparison: Cohort 1: Nivolumab; Null hypothesis is the change in CD8+ cell density is not significantly different from zero; Test type: Superiority; p = 0.08, Wilcoxon Signed-Rank Test
Statistical Analysis 2: Comparison: Cohort 2: Nivolumab/Lirilumab; Test type: Superiority; p = 0.002, Wilcoxon Signed-Rank Test

6. Secondary Outcome: Percentage Change in CD8+ TIL Density
Description: CD8+ TIL density was measured at baseline(TURBT) and radical cystectomy after treatment. The change in CD8+ TIL density from pre-treatment Transurethral Resection of Bladder Tumor (TURBT) to post-treatment Radical Cystectomy (RC) tissues separately in patients treated with nivolumab or combination of nivolumab/liriluma. Each individual patient's percent change was defined as [(Cystectomy TIL Density)-(TURBT TIL Density)] / (TURBT TIL Density) x 100
Time Frame: The outcome was measured from pre-treatment Transurethral Resection of Bladder Tumor (TURBT) to Radical Cystectomy (RC), up to 6 months.TURBT was scheduled 10 weeks at most before the treatment. RC was scheduled within 6 weeks after the last treatment.
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab
Number analyzed (Participants) | 12 | 28
percentage of change | 0.8 [-0.7 to 49.2] | 1.1 [-0.8 to 12.1]
Statistical Analysis 1: Comparison: Cohort 1: Nivolumab vs Cohort 2: Nivolumab/Lirilumab; Test type: Superiority; p = 0.88, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: Participants were followed for AE from the first treatment to 100 days after their last dose of neoadjuvant therapy.
Description: The AEs removed are those do not meet the AE definition. The change of data reported is due to the fact that the AE data have undergone further data cleaning/data management. The result we provide at this time is after the data cleaning.
Arm/Group | Cohort 1: Nivolumab | Cohort 2: Nivolumab/Lirilumab
All-Cause Mortality (participants affected / at risk) | 3/13 | 6/29
Serious Adverse Events (participants affected / at risk) | 3/13 | 6/29
Other Adverse Events (participants affected / at risk) | 12/13 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Nivolumab (N=13) | Cohort 2: Nivolumab/Lirilumab (N=29)
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Nivolumab (N=13) | Cohort 2: Nivolumab/Lirilumab (N=29)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 4
Proctalgia (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 3 | 4
Localised oedema (General disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3
Stoma site pain (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 4
Chills (General disorders) | 0 | 9
Pyrexia (General disorders) | 0 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Vaginal discharge (Reproductive system and breast disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT03532451/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03532451/SAP_001.pdf